CLINICAL TRIAL: NCT01344876
Title: A Dose-escalation Trial to Investigate the Safety and Tolerability of OPB-51602 in Patients With Relapsed or Refractory Hematologic Malignancies (Phase 1)
Brief Title: Phase I Study of OPB-51602 in Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 266-10-001; JapicCTI-111478 (Other: JAPIC)
Record Dates: First submitted 2011-04-26; First posted 2011-04-29 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Myeloma; Non-Hodgkin Lymphoma; Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Chronic Myeloid Leukemia
Keywords: multiple myeloma [MM]; non-Hodgkin lymphoma [NHL]; acute myeloid leukemia [AML]; acute lymphoid leukemia [ALL]; chronic myeloid leukemia [CML]
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPB-51602 (Experimental): OPB-51602 1, 2, 4 and 6 mg/day oral once daily (QD) in a 4 week cycle
  Interventions: Drug: OPB-51602

INTERVENTIONS:
Drug: OPB-51602 — once daily during the treatment period

SUMMARY:
To determine the maximum tolerated dose (MTD) of OPB-51602

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of MM, NHL, AML, ALL or CML.
2. Patients who are responsive or have relapsed following standard treatment
3. Patients capable of providing written informed consent
4. Japanese patients age 20 to 75 years (inclusive) at time of informed consent
5. ECOG performance status score of 0-1
6. Life expectancy of at least 3 months
7. Adequate vital organ function
8. Patients who, together with their partner, are willing and capable of using an appropriate method of contraception throughout the trial period and until at least 12 weeks after final IMP administration

Exclusion Criteria:

1. Patients with other primary malignant tumors
2. Symptomatic CNS involvement
3. Ongoing or active infection, or complication that is not controllable by medication or other means
4. Complication of uncontrolled cardiac disease
5. Female patients who are pregnant, possibly pregnant, or lactating, or who wish to become pregnant during the study period
6. Patients who have received another study drug, or who have received chemotherapy, immunotherapy, cytokine therapy, surgery, or radiotherapy for treatment of the primary disease, within 4 weeks prior to enrollment

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Nagoya
  - Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- OPB-51602: 1mg/Day: OPB-51602: 1, 2, 3,4 and 6 mg/day oral once daily (QD) in a 4 week cycle
- OPB-51602: 2mg/Day; OPB-51602: 3mg/Day; OPB-51602: 4mg/Day; OPB-51602: 6mg/Day: OPB-51602: 1, 2, 3, 4 and 6 mg/day oral once daily (QD) in a 4 week cycle
Period: Overall Study
Arm/Group | OPB-51602: 1mg/Day | OPB-51602: 2mg/Day | OPB-51602: 3mg/Day | OPB-51602: 4mg/Day | OPB-51602: 6mg/Day
Started | 4 | 3 | 4 | 6 | 3
Completed | 3 | 3 | 3 | 3 | 2
Not Completed | 1 | 0 | 1 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Definite progression of primary disease | 1 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- OPB-51602: OPB-51602: 1, 2, 3, 4 and 6 mg/day oral once daily (QD) in a 4 week cycle
  OPB-51602: once daily during the treatment period
Arm/Group | OPB-51602
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  Japan | 20

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Treatment Emergent Adverse Events
Description: Treatment emergent adverse events observed during outcome measure time frame. A Treatment Emergent Adverse Event was defined as an AE occurring after the start of IMP administration.
Time Frame: From first study medication to on Day 31 (after repeated 28 days medication from Day 4 to 31)
Population: Safety population No statistical analysis provided for Subjects With Treatment Emergent Adverse Events.
Measure: Number; unit: participants
Arm/Group | OPB-51602
Number analyzed (Participants) | 20
participants | 20

2. Secondary Outcome: Treatment Response
Description: Assessment of the treatment response was evaluated according to internationally recognized response criteria for multiple myeloma, non-Hodgkin's lymphoma, acute myeloid leukemia, chronic myeloid leukemia.
  "Response" was defined as at least partial response or partial remission (PR) according to the criteria for efficacy assessment.
Time Frame: From first dose of study medication to withdrawal examination
Population: Efficacy population included all treated subjects who had received at least 1 dose of study drug.
  No statistical analysis provided for treatment response.
Measure: Number; unit: participants
Arm/Group | OPB-51602
Number analyzed (Participants) | 20
participants | 0

3. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLT was defined as adverse events occurring during Cycle 1 and: (1) Grade 3 or higher nausea, vomiting, or diarrhea despite the use of anti-emetic or antidiarrheal drugs, (2) Grade 3 or higher non-hematologic toxicity, excluding alopecia, (3) AEs requiring interruption of the IMP for a total of 8 days or longer, (4) Grade 4 neutropenia lasting ≥ 8 days (not applicable for leukemia), (5) Grade 3 or higher febrile neutropenia or infection due to neutropenia (not applicable for leukemia), (6) Grade 4 thrombocytopenia or Grade 3 thrombocytopenia requiring platelet transfusion (not applicable for leukemia).
Time Frame: From first study medication to on Day 31 (after repeated 28 days medication from Day 4 to 31)
Population: DLT evaluated subjects who had achieved ≧75% study drug compliance during a 4-week (28-day) treatment period starting from Day 4. No statistical analysis provided for Subjects With DLTs.
Measure: Number; unit: participants
Groups:
- OPB-51602 1m/Day; OPB-51602 2mg/Day; OPB-51602 3mg/Day; OPB-51602 4mg/Day; OPB-51602 6mg/Day: OPB-51602: 1, 2, 3, 4 and 6 mg/day oral once daily (QD) in a 4 week cycle
Arm/Group | OPB-51602 1m/Day | OPB-51602 2mg/Day | OPB-51602 3mg/Day | OPB-51602 4mg/Day | OPB-51602 6mg/Day
Number analyzed (Participants) | 4 | 3 | 4 | 6 | 3
participants | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study medication to 30 days after last dose of study medication.
Groups:
- OPB-51602 1mg/Day; OPB-51602 2mg/Day; OPB-51602 3mg/Day; OPB-51602 4mg/Day; OPB-51602 6mg/Day: OPB-51602: 1, 2, 3, 4 and 6 mg/day oral once daily (QD) in a 4 week cycle
Arm/Group | OPB-51602 1mg/Day | OPB-51602 2mg/Day | OPB-51602 3mg/Day | OPB-51602 4mg/Day | OPB-51602 6mg/Day
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 2/4 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPB-51602 1mg/Day (N=4) | OPB-51602 2mg/Day (N=3) | OPB-51602 3mg/Day (N=4) | OPB-51602 4mg/Day (N=6) | OPB-51602 6mg/Day (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPB-51602 1mg/Day (N=4) | OPB-51602 2mg/Day (N=3) | OPB-51602 3mg/Day (N=4) | OPB-51602 4mg/Day (N=6) | OPB-51602 6mg/Day (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (2) | 2 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (7) | 1 (2) | 4 (5) | 2 (2) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 3 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 3 (3)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (5)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 4 (6) | 2 (3)
White blood cell count decreased (Investigations) | 2 (2) | 1 (2) | 1 (1) | 3 (4) | 2 (4)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (3)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 2 (2) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No